CLINICAL TRIAL: NCT04898582
Title: A Split-face Study Assessing the Clinical Benefit, Tolerability and Subject Satisfaction of M89PB in Subjects With Rosacea Associated With Erythema and Sensitive Skin
Brief Title: Clinical Benefit of M89PB in Subjects With Rosacea Associated With Erythema and Sensitive Skin
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Institute of Skin and Product Evaluation, Italy (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: E11UE14UE16UT17CS14CSSSB
Record Dates: First submitted 2021-05-12; First posted 2021-05-24 (Actual); Last update posted 2021-05-24 (Actual); Status verified 2021-05

CONDITIONS: Rosacea; Sensitive Skin
MeSH Terms: conditions — Rosacea

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 20 women 20-60 years old with sensitive skin and persistent centrofacial erythema of rosacea (Other): The subjects applied the product M89 Probiotic Fractions on half a face, twice a day, in the morning and in the evening, for 30 days. They put two drops of the product in the palm of their hand and gently massage with their fingertips on half face. The face skin had to be cleaned and dried before the application of the product. The subjects used their standard skin care product on the side of the face not treated with M89 Probiotic Fractions. The subjects were allowed to use their habitual foundation and makeup products on the whole face.
  The side of application of the product M89 Probiotic Fractions (right or left side of the face) was randomized among the subjects.
  The assignment of subject number and subsequent placement on the randomization chart were made in order of appearance at the study centre on the first day.
  Interventions: Other: Mineral 89 Probiotic Fractions

INTERVENTIONS:
Other: Mineral 89 Probiotic Fractions — The subjects applied the product M89 Probiotic Fractions on half a face, twice a day, in the morning and in the evening, for 30 days. They put two drops of the product in the palm of their hand and gently massage with their fingertips on half face. The face skin had to be cleaned and dried before the application of the product. The subjects used their standard skin care product on the side of the face not treated with M89 Probiotic Fractions
  Other Names: Vichy

SUMMARY:
The aim of the study is to assess the efficacy of the product M89 probiotic fractions in improving the symptoms of rosacea patients with sensitive skin after 30 days of treatment, in comparison with an area treated with the habitual skin care product.

20 women with sensitive skin (positive reaction to stinging test), suffering from persistent centrofacial erythema of rosacea with no more than 3 papules and pustules apply the product on half a face, twice a day, for 30 days. The subjects use their habitual skin care product on the other side of the face.

The product efficacy is supported by significant improvements in the mean basal values of the following instrumental parameters: skin hydration (increase), trans-epidermal water loss (decrease), skin erythema (a* parameter decrease).

The efficacy and the tolerability of the product is also showed by a visual clinical assessment of the face skin conditions and by stinging test. Digital images of the face of the subjects were also taken at each control time.

Furthermore, the volunteers express their judgement on the efficacy and the pleasantness of the product by means of a self-assessment questionnaire.

DETAILED DESCRIPTION:
The test was carried out in a temperature and humidity-controlled room (24 ± 2 °C; 50 ± 10 % r.h.).

20 female subjects, between 20 and 60 years old, phototype I-IV according to Fitzpatrick skin type classification, with sensitive skin (positive reaction to stinging test) and suffering from persistent centrofacial erythema of rosacea with no more than 3 papules and pustules were selected for the study.

Volunteers were asked not to wash their face for at least 2 hours before performing the assessments and not to apply any products on the face for 12 hours before the basal visit.

The subjects were recruited for the study if they showed a positive response to stinging test performed with the application of a solution at 15% lactic acid on the nasolabial folds.

The volunteers rated the burning/stinging/itching/painful sensations perceived on each nasolabial fold after 2.5 and 5 minutes from the application, on the basis of the following scale: 0=no burning/stinging/itching/painful sensation; 1=mild burning/stinging/itching/painful sensation; 2=moderate burning/stinging/itching/painful sensation; 3=severe burning/stinging/itching/painful sensation.

If the sum of the score of the two time points was ≥ 3 for each nasolabial fold, the subject was considered a 'stinger', a subject with sensitive skin and could be selected for the test.

The selected subjects filled in a questionnaire on sensitive skin. The subjects applied the product M89 Probiotic Fractions on half a face, twice a day, in the morning and in the evening, for 30 days. They put two drops of the product in the palm of their hand and gently massage with their fingertips on half face. The face skin had to be cleaned and dried before the application of the product. The subjects used their standard skin care product on the side of the face not treated with M89 Probiotic Fractions. The subjects were allowed to use their habitual foundation and makeup products on the whole face.

The side of application of the product M89 Probiotic Fractions (right or left side of the face) was randomized among the subjects.

The assignment of subject number and subsequent placement on the randomization chart were made in order of appearance at the study centre on the first day.

The following evaluations were performed at the baseline, after 15 days and/or after 30 days of treatment:

Instrumental Evaluations: baseline, after 15 days and after 30 days of treatment:

* skin hydration by Corneometer CM825
* trans-epidermal water loss (TEWL) by Tewameter TM 300 MDD 4
* skin erythema by Chromameter CR400

The measurements were performed on the cheeks, on the same location at each control time.

Digital images of the face of the subjects were also taken by means of Fotofinder Dermoscope Ver. 2.0.

Clinical Evaluation: baseline, after 15 days and after 30 days of treatment

A visual clinical evaluation of each side of the face was performed by the technician related to:

* erythema
* desquamation
* number of papules and pustules (visual count)

The subjects were asked to refer about skin tightness, skin dryness, burning, itching, stinging sensations perceived on each side of the face answering to the following questions:

Skin tightness: Do you feel skin tightness? Skin dryness: Does your skin feel dry? Burning sensation: Do you suffer from burning sensation of your skin? Itching sensation: Do you suffer from itching sensation of your skin? Stinging sensation: Do you suffer from stinging/tingling sensation of your skin? The parameters erythema, desquamation, skin tightness, skin dryness, burning, itching and stinging were scored according to a 0-10 scale.

Stinging Test: baseline, after 15 days and after 30 days of treatment

A solution at 15% lactic acid was applied on the nasolabial folds of each subject. The volunteers rated the burning/stinging/itching/pain sensations perceived on each nasolabial fold after 2.5 and 5 minutes from the application, on the basis of the following scale:

0=no burning/stinging/itching/painful sensation;

1. mild burning/stinging/itching/painful sensation;
2. moderate burning/stinging/itching/painful sensation;
3. severe burning/stinging/itching/painful sensation.

Standardized Skin Surface Biopsy technique (SSSB): after 30 days of treatment The face of the volunteers was cleaned with ether to remove traces of sebum. Then a drop (about 0.05 ml) of cyanoacrylate glue was homogeneously applied to an area of 1 cm 2 at one end of a microscope slide. Then the slide (SSSB 1) was put against one cheek. The slide was left in place until the cyanoacrylate changed in consistency and then gently removed. A second SSSB (SSSB 2) was performed at the same site immediately after the first. The procedure was repeated on the other cheek in order to collect slides related to both the areas (treated with M89 and with the habitual skin care product). The SSSB 2 were analyzed with a microscope (x40) and the Demodex density (number of Demodex in 1 cm2) was determined for each slide.

Satisfaction questionnaire: after 15 days and after 30 days of treatment The subjects expressed their opinion on the efficacy and the pleasantness of the product by filling in a questionnaire referred to the side of the face treated with M89 Probiotic Fractions.

ELIGIBILITY:
Inclusion Criteria:

* Caucasian subjects of female sex, 20-60 years old, phototype I-IV according to Fitzpatrick skin type classification and in good general health.
* Subjects with sensitive skin (positive reaction to stinging test, score ≥ 3).
* Subjects suffering from persistent centrofacial erythema of rosacea with no more than 3 papules and pustules.
* Subjects able to follow all study directions and willing to commit to all follow-up visits for the duration of the study.
* Subjects who have completed the written informed consent process.
* Subjects who avoid the exposure to UV radiation and the use of tanning beds for the duration of the study.

Exclusion Criteria:

* Pregnant or nursing females.
* Subjects with Rosacea and more than 3 papules or pustules.
* Subjects who are taking topical or systemic drugs that could affect the results of the test (immunosuppressants, anti-inflammatory agents, corticosteroids, etc.).
* Subjects with a change in contraception.
* Subjects showing systemic diseases or skin disorders (such as eczema, psoriasis, severe acne, etc.) that may affect the evaluation of the test articles or increase risk to the subject.
* Subjects who have used treatments for rosacea (either topical and/or systemic) within a period of 30 days prior to admission in this study.
* Subjects who have been involved in another clinical investigation with comparable purposes within a period of 30 days prior to admission in this study.

Ages: 20 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2021-05-18 (Actual); Primary Completion 2021-05-18 (Actual); Study Completion 2021-05-18 (Estimated)

PRIMARY OUTCOMES:
skin hydration (change of skin hydration from baseline is being assessed at 15 and 30 days) | baseline, 15 days and 30 days of treatment
  Corneometer CM825
  Corneometer CM 825 measures the skin hydration. The instrument is based on the physical principle of capacitance. The corneometric values increase with increasing hydration of the stratum corneum. The efficacy of the product in improving skin hydration is evidenced by an increase of the average corneometric values.
Trans-epidermal water loss - TEWL (change of TEWL from baseline is being assessed at 15 and 30 days) | baseline, 15 days and 30 days of treatment
  Tewameter TM 300 MDD 4
  Tewameter TM 300 measures the trans-epidermal water loss (TEWL) on the base of Fick's diffusion formula. TEWL values reflects the skin barrier function.
  TEWL (Trans-epidermal Water Loss) expressed in g/h m2 increases with increasing impairment of skin barrier function.
skin erythema - a* parameter (change of skin erythema from baseline is being assessed at 15 and 30 days) | baseline, 15 days and 30 days of treatment
  Chromameter CR400
  Chromameter is a portable dual channel, reflecting colorimeter with incorporated microcomputer, liquid crystals display and Xenon light source in the measuring head. The measuring head surface is 8 mm in diameter.
  The colour rating system is CIE system L*a*b*:
  In the present study only the values related to the a* parameter were taken into consideration as index of skin redness/erythema.
  a* value linearly increases with increasing of the intensity of the erythema.
Stinging test (change of stinging test clinical scores from baseline is being assessed at 15 and 30 days) | baseline, 15 days and 30 days of treatment
  A solution at 15% lactic acid was applied on the nasolabial folds of each subject. The volunteers rated the burning/stinging/itching/pain sensations perceived on each nasolabial fold after 2.5 and 5 minutes from the application, on the basis of the following scale:
  0=no burning/stinging/itching/painful sensation;
  1. mild burning/stinging/itching/painful sensation;
  2. moderate burning/stinging/itching/painful sensation;
  3. severe burning/stinging/itching/painful sensation.
Clinical evaluation (change of clinical scores from baseline is being assessed at 15 and 30 days) | baseline, 15 days and 30 days of treatment
  A visual clinical evaluation of each side of the face was performed by the technician related to:
  * erythema
  * desquamation
  * number of papules and pustules (visual count)
  The subjects were asked to refer about skin tightness, skin dryness, burning, itching, stinging sensations perceived on each side of the face answering to the following questions:
  Skin tightness: Do you feel skin tightness? Skin dryness: Does your skin feel dry? Burning sensation: Do you suffer from burning sensation of your skin? Itching sensation: Do you suffer from itching sensation of your skin? Stinging sensation: Do you suffer from stinging/tingling sensation of your skin?
  The parameters erythema, desquamation, skin tightness, skin dryness, burning, itching and stinging were scored according to the following 0-10 scale:
  0 1 2 3 4 5 6 7 8 9 10 Not at all Extremely
Standardized Skin Surface Biopsy (SSSB) | 30 days of treatment
  The face of the volunteers was cleaned with ether to remove traces of sebum. Then a drop (about 0.05 ml) of cyanoacrylate glue was homogeneously applied to an area of 1 cm 2 at one end of a microscope slide. Then the slide (SSSB 1) was put against one cheek. The slide was left in place until the cyanoacrylate changed in consistency and then gently removed. A second SSSB (SSSB 2) was performed at the same site immediately after the first. The procedure was repeated on the other cheek in order to collect slides related to both the areas (treated with M89 and with the habitual skin care product). The SSSB 2 were analyzed with a microscope (x40) and the Demodex density (number of Demodex in 1 cm2) was determined for each slide.
Digital Images (change is being assessed) | baseline, 15 days and 30 days of treatment
  Digital images of the face of the subjects were also taken by means of Fotofinder Dermoscope Ver. 2.0.

SECONDARY OUTCOMES:
Satisfaction Questionnaire | 15 days and 30 days of treatment
  The subjects expressed their opinion on the efficacy and the pleasantness of the product by filling in a questionnaire referred to the side of the face treated with M89 Probiotic Fractions.

CONTACTS AND LOCATIONS:
Overall Officials: Claudia Cartigliani, Principal Investigator — ISPE srl
Locations (1):
- ISPE srl, Milan, MI, Italy

IPD SHARING:
Plan to Share IPD: No